CLINICAL TRIAL: NCT01083966
Title: Phase I Trial of Super-Selective Intraarterial Cerebral Infusion of Bevacizumab (Avastin) for Treatment of Vestibular Schwannoma (Acoustic Neuroma)
Brief Title: Super-Selective Intraarterial Cerebral Infusion of Bevacizumab (Avastin) for Treatment of Vestibular Schwannoma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Feinstein Institute for Medical Research (Other); Hofstra North Shore (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Professor, Feinstein Institute for Medical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0912010765
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Vestibular Schwannoma
Keywords: Vestibular; Schwannoma; earing-loss; brain-tumor; Acoustic; Neuroma
MeSH Terms: conditions — Neuroma, Acoustic; Neurilemmoma; Brain Neoplasms; Neuroma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin (Experimental): IA Avastin
  Interventions: Drug: Bevacizumab (Avastin)

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — Super-Selective Intraarterial Intracranial Infusion of Bevacizumab in Vestibular Schwannoma
  This phase I clinical research trial will test the hypothesis that Bevacizumab can be safely used by direct intracranial superselective intraarterial infusion up to a dose of 10mg/kg to ultimately enhance survival and hearing function of patients with VS
  Other Names: Avastin

SUMMARY:
A recent study by Plotkin et al. showed that bevacizumab (Avastin) treatment was followed by clinically meaningful hearing improvement, tumor-volume reduction, or both in some, but not all, patients with Vestibular Schwannoma (VS) who were at risk for complete hearing loss or brain-stem compression from growing VS. Because of the promising results in preliminary studies of Bevacizumab and because of significant experience with the safety of the dosages proposed in this study, this study will offer a safe treatment for patients with VS. Therefore, this phase I clinical research trial will test the hypothesis that Bevacizumab can be safely used by direct intracranial superselective intraarterial infusion up to a dose of 10mg/kg to ultimately enhance survival and hearing function of patients with VS.

DETAILED DESCRIPTION:
Newer techniques in interventional neuroradiology have allowed for a more selective delivery of catheters higher up into the arterial tree where agents such as chemotherapies, can be delivered without the risk of adverse affects such as blindness. In fact, studies here at Cornell have developed very new and exciting super selective intraarterial delivery treatment for Retinoblastoma and Malignant Glioma brain tumors with little toxicity. Therefore, this trial will ask one simple question: Is it safe to deliver a first dose of Avastin intraarterially using these super selective delivery techniques instead of the standard intravenous route of administration? This should not only increase the amount of drug that gets to the VS but also spare them of any adverse effects from a less selective delivery. During that single dose of intraarterial Avastin, they will also receive a dose of mannitol that opens up the blood brain barrier to improve delivery of the agent to the tumor. After that single dose of Mannitol and Avastin intraarterially, the patient will be evaluated for 4 weeks to assess for toxicity. If no toxicity, then the will go on and get MRI of the brain every two months to assess for response up to 12 months. After this, the subject is done with the "experimental" aspects of the protocol. This is a Phase I trial that is designed to test the safety of the single dose intraarterial delivery of Avastin and Mannitol,.

To summarize:

Current Standard of Care: Surgery or radiosurgery: IV Avastin

Experimental portion of this proposal:

Day 0: Intraarterial Avastin single dose (starting at 2mg/kg and up to 10mg/kg) after Mannitol to open the blood brain barrier Day 28 (and every two months thereafter): MRI brain with contrast

Therefore the experimental aspects of this treatment plan will include:

1. Subjects will first be treated with Mannitol prior to chemotherapy infusion (Mannitol 25%; 3-10 mL/s for 30seconds) in order to disrupt the blood brain barrier. This technique has been used in several thousand patients in previous studies for the IA delivery of chemotherapy for malignant glioma.
2. To add a single intraarterial delivery (SIACI) of the Avastin with VS.
3. The dose escalation algorithm is as follows: We will use a single intracranial superselective intraarterial infusion of Avastin, starting at a dose of 2mg/kg in the first three patients. Assuming no dose limiting toxicity during the first 28 days after IA infusion, an MRI of the brain will be performed. The doses will be escalated to 4,6,8 and finally 10mg/kg in this Phase I trial.

Inclusion criteria Include: Males or females, >=18 years of age, with documented Radiologic or histologic diagnosis of VS

Both hematologic and non-hematologic toxicity will be determined and scored according to the NCI Common Toxicity Criteria (version 3.0). Monitoring will be conducted by post procedure history, neurological and physical examinations together with serial blood counts, prothrombin time (PT), partial thromboplastin time (PTT) and chemistries.

Response will be evaluated after 4 weeks via a MRI with the injection of contrast. The following will be evaluated every cycle, and then during follow-up: neurological examination, physical examination, performance status, laboratory parameters and review of adverse reactions. Contrast enhanced MRI (MRI with gadolinium is the preferable imaging study. The following subjects will be taken off protocol: those with progressive disease; those who experience dose-limiting toxicity (DLT). Follow-up will continue until disease progression or death. Survival will be measured from the time of the first dose of IA Avastin® (given at the start of each treatment cycle).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of >= 18 years of age.
* Patients with a documented diagnosis of unilateral or bilateral VS based on MRI and who have evidence of progressive vestibular schwannomas, and are considered poor candidates for surgery and radiation therapy or declined these treatments.
* Patients must have a Karnofsky performance status >=60% (or the equivalent ECOG level of 0-2) (see Appendix A; Performance Status Evaluation) and an expected survival of >= three months.
* No chemotherapy for two weeks prior to treatment under this research protocol and no external beam radiation for two weeks prior to treatment under this research protocol.
* Patients must have adequate hematologic reserve with WBC>=3000/mm3, absolute neutrophils >=1500/mm3 and platelets >=100,000/ mm3. Patients who are on Coumadin must have a platelet count of >=150,000/ mm3.
* Pre-enrollment chemistry parameters must show: bilirubin< 1.5X the institutional upper limit of normal (IUNL); AST or ALT< 2.5X IUNL and creatinine < 1.5X IUNL.
* Pre-enrollment coagulation parameters (PT and PTT) must be <1.5X the IUNL.
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.

Exclusion Criteria:

* Previous treatment with Avastin®.
* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring including MRI with gadolinium.
* Surgery (including open biopsy), significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during study treatment.
* Current or recent (within 10 days of Avastin) use of aspirin (> 325 mg/day), full dose (i.e., therapeutic dose) of oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes. Prophylactic use of anticoagulants is allowed (e.g., warfarin (1 mg qd) for catheter prophylaxis, and prophylactic low molecular-weight heparin (i.e., enoxaparin [(40mg QD0]).
* History or evidence of inherited bleeding diathesis or coagulopathy with a risk of bleeding.
* Inadequately controlled hypertension (blood pressure: systolic > 150 mmHg and/or diastolic > 100 mmHg).
* Patients with baseline urine dipstick for proteinuria > 2+ must undergo a 24-hours urine collection and must demonstrate ≤ 1 g of protein in 24 hours.
* Clinically significant (i.e., active) cardiovascular disease (e.g., cerebrovascular accident or myocardial infarction within 6 months prior to randomization),unstable angina, congestive heart failure (NYHA Class ≥ II), or serious cardiac arrhythmia that is uncontrolled by medication or may interfere with administration of study treatment.
* Serious non-healing sound, active peptic ulcer, or untreated bone fracture.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of enrollment.
* Known hypersensitivity to Avastin or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose. | 1 month post procedure

SECONDARY OUTCOMES:
Composite overall response rate | 2 years
Six-month progression-free survival (PFS) | 6 months
Hearing response will be assessed in eligible patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States